CLINICAL TRIAL: NCT02456480
Title: A Randomized, Double-blind, Placebo Controlled Study to Assess the Pharmacodynamics, Safety/Tolerability and Efficacy of Omiganan in Patients With Mild to Moderate Atopic Dermatitis
Brief Title: Pharmacodynamics of Omiganan (CLS001) in Patients With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maruho Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLS001-CO-PR-008; 2014-003689-26 (EudraCT Number)
Record Dates: First submitted 2015-05-01; First posted 2015-05-28 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CLS001 topical gel, 2.5% (Experimental)
  Interventions: Drug: CLS001
- CLS001 topical gel 1% (Experimental)
  Interventions: Drug: CLS001
- Vehicle gel (Placebo Comparator)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: CLS001 — topical gel
  Arms: CLS001 topical gel 1%; CLS001 topical gel, 2.5%
Drug: Vehicle — topical gel
  Arms: Vehicle gel

SUMMARY:
To assess the pharmacodynamics, safety/tolerability, and efficacy of omiganan in patients with mild to moderate atopic dermatitis (AD).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects with mild to moderate AD 18 to 65 years of age, inclusive.
2. AD diagnosed by physician / medical specialist and that has been (intermittently) present for at least 1 year
3. Able to participate and willing to give written informed consent and to comply with the study restrictions.

Exclusion Criteria:

1. Have any current and / or recurrent clinically significant skin condition in the treatment area other than AD.
2. Any confirmed, active significant allergic reactions (urticaria or anaphylaxis) including allergic reactions against any drug, multiple drug allergies or (ingredients of) emollients.
3. Participation in an investigational drug or device study within 3 months prior to screening or more than 4 times a year.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-05; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamic (Local punch biopsy of a target lesion pre-dose and post treatment for the change in biomarkers including IL, filaggrin, TLR, IgE, IFN, and microbiome of the skin lesion) | 42 Days
  Local punch biopsy of a target lesion pre-dose and post treatment for the change in biomarkers including IL, filaggrin, TLR, IgE, IFN, and microbiome of the skin lesion
Clinical assessment (Change in patient symptoms over time using pruritis VAS) | 42 Days
  Change in patient symptoms over time using pruritis VAS
Clinical Assessment (Change in lesion size over time) | 42 Days
  Change in lesion size over time
Clinical assessment (Change in patient SCORAD scale score over time) | 42 Days
  Change in patient SCORAD scale score over time

SECONDARY OUTCOMES:
Safety Assessment (Adverse events) | 42 days
  Adverse events will be collected throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: J. (Koos) Burggraaf, MD, PhD, Principal Investigator — Centre for Human Drug Research
Locations (1):
- Centre for Human Drug Research, Zernikedreef 8, Netherlands

REFERENCES:
- [Derived] Niemeyer-van der Kolk T, van der Wall H, Hogendoorn GK, Rijneveld R, Luijten S, van Alewijk DCJG, van den Munckhof EHA, de Kam ML, Feiss GL, Prens EP, Burggraaf J, Rissmann R, van Doorn MBA. Pharmacodynamic Effects of Topical Omiganan in Patients With Mild to Moderate Atopic Dermatitis in a Randomized, Placebo-Controlled, Phase II Trial. Clin Transl Sci. 2020 Sep;13(5):994-1003. doi: 10.1111/cts.12792. Epub 2020 May 1. PMID 32315497